CLINICAL TRIAL: NCT00681460
Title: Effects of Insulin and/or Metformin Treatment on Perinatal Outcome and Metabolic Parameters in Women With Gestational Diabetes Mellitus: Prospective Randomized Trial.
Brief Title: Metformin in Gestational Diabetes Mellitus
Acronym: MetGDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: K. Marcinkowski University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Agnieszka Zawiejska, MD, PhD, Department of Obstetrics and Women's Diseases, Senior Lecturer, K. Marcinkowski University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUMS 705/07
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes, Gestational; Insulin Resistance
Keywords: gestational diabetes; birth weight; fetal growth; insulin resistance; oxidative stress; inflammatory reaction; Fetal Development
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance; Birth Weight; Inflammation | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): gestational diabetes, insulin therapy
  Interventions: Drug: human recombined insulin
- 2 (Experimental): gestational diabetes, metformin therapy
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: human recombined insulin — multiple injections protocol (functional intensive insulin therapy), variable doses following dietary conditions and current metabolic status
  Arms: 1
Drug: metformin — pills given orally twice up to three times a day, a total daily dosage 1000-2400 mg
  Arms: 2

SUMMARY:
Gestational diabetes (GDM) is a condition that manifests as high blood sugar levels (hyperglycemia) during pregnancy in previously healthy women. It develops as a result of increased maternal body's resistance to insulin - a major hormone that allows for utilisation of glucose (sugar taken in with food) within cells. It was found out that GDM occurs more frequently in overweight women but also in women with a history of certain conditions such as polycystic ovary syndrome (PCOS). Usually, GDM disappears after pregnancy is completed but it is associated with some serious hazards for women and her unborn child, if untreated properly. Diet is a first-choice treatment but sometimes insulin therapy must be initiated if keeping a diet alone is not enough to maintain blood sugar within recommended values. Insulin therapy is effective but it requires several injections during each day and insulin is a strong acting hypoglycemic agent that may induce rapid falls in blood sugar, also dangerous for mother and unborn child.

In the investigators study, the investigators would like to investigate if metformin that is a commonly used hypoglycemic drug can be effectively used for GDM treatment. Metformin has been used successfully for a long time to treat type 2 diabetes mellitus and PCOS and, according to current data, it is not dangerous neither for mother nor for baby when used during gestation.

ELIGIBILITY:
Inclusion Criteria:

* diabetes diagnosed during pregnancy
* single pregnancy
* ineffective diet therapy

Exclusion Criteria:

* pregestational diabetes
* fetal malformation
* multiple pregnancy
* contraindications to metformin therapy (liver or kidney disease)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-05; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
newborn weight | first hour of life

SECONDARY OUTCOMES:
parameters of metabolic control in mother and newborn, insulin resistance, inflammatory reaction, oxidative stress, fetal growth, | during pregnancy and up to twelve hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Brazert, MD.PhD.prof, Study Chair — K Marcinkowski University of Med Sciences, Poznan, Poland; Antoni J Duleba, MD.prof, Study Director — University of California at Davis, Sacramento, CA, USA
Locations (1):
- Div of Obstetrics and Women's Diseases, Dept of Obstetrics and Gynecology, K Marcinkowski Univ of Med Sciences, Poznan, Poland